CLINICAL TRIAL: NCT03093181
Title: A Randomized, Parallel-group, Evaluator-blind, No-treatment and Positive Controlled, Single-site, Proof of Concept Clinical Study to Evaluate the Cosmetic Benefit Provided by 8 Weeks of Twice-daily Topical Application of a Developmental Moisturizing Cream With Niacinamide in Healthy Subjects With Sensitive, Oily, Blemish-prone Skin
Brief Title: A Study to Evaluate of Cosmetic Benefit of a Moisturising Cream in People With Blemish Prone Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 207196
Record Dates: First submitted 2017-03-24; First posted 2017-03-28 (Actual); Results first posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Skin Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No treatment and Standard cleanser (Placebo Comparator): Participants randomised to the no treatment regimen will use the standard cleanser (only) twice a day (morning and night). Morning and evening applications should be separated by at least 8 hours.
  Interventions: Other: Washout / Standard Cleanser
- Test product and Standard cleanser (Experimental): Participants randomised to test product regimen will be instructed to use the standard cleanser and test product twice a day (morning and night). Morning and evening applications should be separated by at least 8 hours. Participants will be instructed to apply the test product cream immediately after cleansing.
  Interventions: Other: Washout / Standard Cleanser; Other: Test product
- Positive control and positive cleanser (Active Comparator): Participants randomised to positive control regimen will be instructed to use the positive cleanser and positive control product twice a day (morning and night). Morning and evening applications should be separated by at least 8 hours. Participants will be instructed to apply the positive control cream immediately after cleansing.
  Interventions: Other: Positive control cleanser; Other: Positive control moisturiser

INTERVENTIONS:
Other: Washout / Standard Cleanser — Participants will apply standard cleanser (Simple Kind to Skin Moisturising Facial Wash) twice daily (morning and night) with at least 8 hours between product applications. Participants will use the standard cleanser in a 5-7 day washout period and during the test phase of the study
  Arms: No treatment and Standard cleanser; Test product and Standard cleanser
Other: Test product — Participants will apply 0.6 gram (g) of Test product (Moisturising Cream with Niacinamide) twice daily (morning and night) with at least 8 hours between product applications. Participants will use the test product during the test phase of the study.
  Arms: Test product and Standard cleanser
Other: Positive control cleanser — Participants will apply positive control cleanser (Neutrogena Visibly Clear Spot Clearing Facial Wash) twice daily (morning and night) with at least 8 hours between product applications. Participants will use the positive control cleanser during the test phase of the study.
  Arms: Positive control and positive cleanser
Other: Positive control moisturiser — Participants will apply 0.6 g of positive control moisturiser (Vivatinell Acnecinamide Gel Cream) twice daily (morning and night) with at least 8 hours between product applications. Participants will use the positive control moisturiser during the test phase of the study.
  Arms: Positive control and positive cleanser

SUMMARY:
This study is designed to evaluate the cosmetic benefit provided by twice daily application of a developmental moisturising cream with niacinamide for 8 weeks in healthy female participants with sensitive, oily, blemish-prone skin.

DETAILED DESCRIPTION:
This study broadly consists of two phases: screening / washout phase (5-7 day) followed by treatment phase (approximately of 8 weeks). Participants will be asked to return to the study site 1 week, 4 weeks and 8 weeks after their randomisation visit for instrumental measurements and clinical assessments.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form
* Good general and mental health with, in the opinion of the investigator or medically qualified designee no clinically significant and relevant abnormalities in medical history or upon physical examination
* Willingness to actively participate in the study and to attend all scheduled visits
* Minimum of 10 and maximum of 25 blemishes (papules and pustules) at Visit 1 and a minimum of 8 blemishes (papules and pustules) at Visit 2
* Fitzpatrick photo-type I-V
* Sebumeter score of >66 µg / cm2 at the forehead
* Females of childbearing potential who are, in the opinion of the investigator, practicing a reliable method of contraception. Adequate contraception is defined as abstinence, oral contraceptive, either combined or progestogen alone OR injectable progestogen OR implants of levonorgestrel OR estrogenic vaginal ring OR percutaneous contraceptive patches OR intrauterine device or intrauterine system OR double barrier method (condom or occlusive cap [diaphragm or cervical vault caps] plus spermicidal agent [foam, gel, film, cream, suppository]) OR male partner sterilization prior to the female participant's entry into the study, and this male is the sole partner for that participant
* Cleanses their face at least once a day

Exclusion Criteria:

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study
* Women who are breast-feeding
* Medical history of using a medicated acne treatment (e.g. Benzoyl Peroxide, Clindamycin, isotretinoin) within the last 12 months
* Change in contraception within the last 3 months
* Active skin disease in the test area
* Medical history of dysplastic nevi or melanoma on the face
* Moles, cysts, tattoos, scars, irritated skin, hairs, etc. at the test area that could influence the investigation
* Systemic therapy with immuno-suppressive drugs (e.g. corticosteroids) and/or antihistamines within 7 days prior to the start of the study and/or throughout the entire course of the study
* Systemic use of anti-microbials within the last month
* Systemic use of over-the-counter (OTC) analgesics or anti-inflammatory drugs 24 hours prior to dosing at the first assessment visit
* One of the following illnesses that might require regular systemic medication: Insulin-dependent diabetes, cancer
* One of the following illnesses if not medicated: Asthma, hypertension
* Medical history of abnormal response to sunlight
* History of mental illness
* Medically diagnosed acne vulgaris, acne conglobate, fulminans, secondary acne (drug induced acne) or any acne requiring systemic or topical treatment
* No aesthetic, cosmetic or dermatological treatment in the treatment area (face) within the last month
* No intense sun exposure, Ultraviolet-treatments or tanning salon visit within the last 2 weeks
* Known or suspected intolerance, allergy or hypersensitivity to study materials (or closely related compounds) or any of their stated ingredients
* History of allergies to cosmetic products or medicated acne treatments
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit
* Previous participation in this study
* Recent history (within the last 5 years) of alcohol or other substance abuse
* An employee of the sponsor or the study site or members of their immediate family

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 157 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2017-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Valinhos, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Santos-Caetano JP, Gfeller CF, Mahalingam H, Thompson M, Moore DJ, Vila R, Doi R, Cargill MR. Cosmetic benefits of a novel biomimetic lamellar formulation containing niacinamide in healthy females with oily, blemish-prone skin in a randomized proof-of-concept study. Int J Cosmet Sci. 2020 Feb;42(1):29-35. doi: 10.1111/ics.12576. Epub 2020 Jan 6. PMID 31461548
- See also: Cosmetic benefits of a novel biomimetic lamellar formulation containing niacinamide in healthy females with oily, blemish-prone skin in a randomised proof-of-concept study. — https://www.ncbi.nlm.nih.gov/pubmed/31461548
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217381&parentIdentifier=207196&attachmentIdentifier=82c32de7-7cba-4b55-8e0e-23f3b181b0c8&fileName=gsk-207196-reporting-and-analysis-plan-redact.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All the participants were recruited from one center in Brazil.
Pre-assignment Details: Out of 205 screened participants,157 participants were enrolled, and 132 participants were randomized. 25 enrolled subjects were not subsequently randomized. Out of 132 randomized participants,1 participant was misallocated to treatment (received "no treatment" instead of "positive control").
Groups:
- Test Product Regimen: Participants randomized to test product regimen used the standard cleanser and test product twice a day (morning and night). Morning and evening applications were separated by at least 8 hours. Participants applied the test product cream immediately after cleansing.
- No Treatment Regimen: Participants randomized to the no treatment regimen used the standard cleanser (only) twice a day (morning and night). Morning and evening applications were separated by at least 8 hours.
- Positive Control Regimen: Participants randomized to positive control regimen used the positive cleanser and positive control product twice a day (morning and night). Morning and evening applications were separated by at least 8 hours. Participants applied the positive control cream immediately after cleansing.
Period: Overall Study
Arm/Group | Test Product Regimen | No Treatment Regimen | Positive Control Regimen
Started | 44 | 44 | 44
Completed | 41 | 42 | 41
Not Completed | 3 | 2 | 3
Not completed — Withdrawal by Subject | 2 | 1 | 2
Not completed — Other (Not specified) | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Other (Protocol violation) | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population(N=132) included all participants who were randomized and received at least 1 dose of study product.1 participant was misallocated to treatment (received "no treatment" instead of "positive control").Total of 45 and 43 participants were included in safety population for "no treatment" and "positive control" respectively.
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Product Regimen | No Treatment Regimen | Positive Control Regimen | Total
Number analyzed (Participants) | 44 | 45 | 43 | 132
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.4 (5.82) | 25.8 (6.05) | 24.8 (5.72) | 25.3 (5.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 45 | 43 | 132
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 5 | 0 | 8
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 14 | 10 | 18 | 42
  White | 27 | 30 | 24 | 81
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Corneometer Values at 8 Hours on Day 1
Description: A blinded, trained and qualified evaluator conducted instrumental measurements of skin moisturization.Measurement of skin moisturization was performed by the electrical capacitance method with a Corneometer CM 865. The measuring principle was based on changes in the capacitance of the measuring head, functioning as a condensator. Between the conductors of the probe an electrical field was built which allows the dielectricity of the stratum corneum to be measured. Because the dielectricity of the skin varies as a function of its water content.The range of hydration level was 0 (as dry as possible)~120 AU (Arbitrary Unit)(most moist possible).Higher Corneometer values are indicative of improved skin moisturization.
Time Frame: At Baseline and Day 1
Population: Intent to treat (ITT, N= 132) population included all participants who were randomized into the study and have at least one post-baseline measurement available.
Measure: Mean (Standard Deviation); unit: Arbitrary Corneometer unit
Arm/Group | Test Product Regimen | No Treatment Regimen | Positive Control Regimen
Number analyzed (Participants) | 44 | 44 | 43
Arbitrary Corneometer unit | 6.14 (6.442) | 2.63 (5.602) | 3.60 (7.860)
Statistical Analysis 1: Comparison: Test Product Regimen vs No Treatment Regimen; Test type: Superiority; p = 0.0128, ANCOVA — From Analysis of covariance (ANCOVA) with treatment main effect, age stratum and baseline as covariates; Least square (LS) mean difference = 3.12, 95% CI 2-sided [0.68 to 5.56] — Difference is first named treatment (test product) minus second named treatment (negative control) such that a positive value favors the first named treatment (test product)
Statistical Analysis 2: Comparison: No Treatment Regimen vs Positive Control Regimen; Test type: Superiority; p = 0.2262, ANCOVA — From ANCOVA with treatment main effect, age stratum and baseline as covariates; LS mean difference = 1.51, 95% CI 2-sided [-0.95 to 3.96] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Corneometer Values at 1 and 3 Hours on Day 1 and at Week 1, 4 and 8
Description: A blinded, trained and qualified evaluator conducted instrumental measurements of skin moisturisation. Measurement of skin moisturisation was performed by the electrical capacitance method with a Corneometer CM 865. The measuring principle was based on changes in the capacitance of the measuring head, functioning as a condensator. Between the conductors of the probe an electrical field was built which allows the dielectricity of the stratum corneum to be measured. Because the dielectricity of the skin varies as a function of its water content. Higher Corneometer values are indicative of improved skin moisturisation.
Time Frame: At Baseline, Day 1, Week 1, 4 and 8
Population: ITT (N= 132) population included all participants who were randomized into the study and have at least one post-baseline measurement available.
Measure: Mean (Standard Deviation); unit: Arbitrary Corneometer unit
Arm/Group | Test Product Regimen | No Treatment Regimen | Positive Control Regimen
Number analyzed (Participants) | 44 | 44 | 44
Arbitrary Corneometer unit
  At 1 hour, Day 1 | 11.52 (8.264) | -3.69 (6.150) | 4.55 (8.055)
  At 3 hour, Day 1 | 9.64 (5.986) | 0.68 (5.029) | 4.33 (7.913)
  At Week 1: number analyzed (Participants) | 44 | 43 | 43
  At Week 1 | 4.39 (10.549) | 0.06 (9.024) | 3.31 (11.027)
  At Week 4: number analyzed (Participants) | 42 | 42 | 41
  At Week 4 | 4.33 (8.935) | 3.16 (7.028) | 1.04 (8.124)
  At Week 8: number analyzed (Participants) | 41 | 42 | 41
  At Week 8 | 7.54 (11.994) | 3.32 (10.059) | 2.51 (12.969)

3. Secondary Outcome: Odds for Logistic Regression Analysis on Improvement Rating of Lay Person Assessment of Polarized and Non-polarized Images Week 8 Compared to Baseline
Description: The baseline and week 8 photographs of all participants were displayed side by side on high resolution, color-calibrated display screen in room with neutral wall colors and standardized lighting and all practical efforts were made to minimize glare. The relative positioning (left and right) of baseline and week 8 photographs were blinded to evaluator and randomized. A technician used randomization schedule to display pair of images to lay evaluator. Lay evaluators judged magnitude of improvement in overall appearance of blemishes using the below criteria: Left=blemishes on left are more obvious than those on the right and Right=blemishes on right are more obvious than those on the left. Layperson ranked both left and right image as follows:1=Better;2=Worse. Odds was calculated from logistic regression including treatment and age stratum effects and exchangeable correlation. Odds=p/(1-p) where p was the probability of event that Week 8 was better than baseline.
Time Frame: At Baseline and Week 8
Population: as for outcome 2
Measure: Number; unit: Odds
Arm/Group | Test Product Regimen | No Treatment Regimen | Positive Control Regimen
Number analyzed (Participants) | 44 | 44 | 44
Odds
  For Polarised Image | 1.84 | 1.00 | 1.04
  For Non-polarised Image | 2.06 | 1.08 | 1.02
Statistical Analysis 1: Comparison: Test Product Regimen vs No Treatment Regimen; Analysis of Lay Person Assessment Polarised Image; Test type: Superiority; p = 0.0243, Odds Ratio; Odds Ratio (OR) = 1.85, 95% CI 2-sided [1.08 to 3.15]
Statistical Analysis 2: Comparison: No Treatment Regimen vs Positive Control Regimen; Analysis of Lay Person Assessment Polarised Image; Test type: Superiority; p = 0.8931, Odds Ratio; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.61 to 1.78]
Statistical Analysis 3: Comparison: Test Product Regimen vs No Treatment Regimen; Analysis of Lay Person Assessment Non-Polarised Image; Test type: Superiority; p = 0.0181, Odds Ratio; Odds Ratio (OR) = 1.90, 95% CI 2-sided [1.12 to 3.25]
Statistical Analysis 4: Comparison: No Treatment Regimen vs Positive Control Regimen; Analysis of Lay Person Assessment Non-Polarised Image; Test type: Superiority; p = 0.8319, Odds Ratio; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.55 to 1.63]

4. Secondary Outcome: ANOVA Analysis on Improvement Rating of Lay Person Assessment of Polarized and Non-polarized Images Week 8 Compared to Baseline
Description: Baseline and Week 8 photographs of all participants were displayed side by side on high resolution, color-calibrated display screen in room with neutral wall colors and standardized lighting with minimized glare. Relative positioning (left and right) of baseline and Week 8 photographs were blinded to evaluator and randomized. Lay evaluators ranked magnitude of improvement in overall appearance of blemishes using below criteria: Left=blemishes on left are more obvious than those on right; Right=blemishes on right are more obvious than those on left. Lay evaluator ranking for each image pair was converted into a numerical score based on whether Baseline or Week 8 image was ranked better:0=Baseline image was better than Week 8 image,1=Week 8 image was better than Baseline image. Minimum score 0 corresponded to all baseline images being better than Week 8 images. Maximum score 1 corresponded to all Week 8 images being better than baseline images. Higher scores indicated better results.
Time Frame: At Baseline and Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Test Product Regimen | No Treatment Regimen | Positive Control Regimen
Number analyzed (Participants) | 44 | 44 | 44
Score on scale
  For Polarised Image | 0.65 (0.048) | 0.50 (0.047) | 0.51 (0.047)
  For Non-polarised Image | 0.67 (0.047) | 0.52 (0.046) | 0.51 (0.047)
Statistical Analysis 1: Comparison: Test Product Regimen vs No Treatment Regimen; Analysis of Lay Person Assessment Polarised Image; Test type: Superiority; p = 0.0279, ANOVA; ANOVA= average rate over all raters including effects of treatment and age stratum; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [0.02 to 0.28]
Statistical Analysis 2: Comparison: No Treatment Regimen vs Positive Control Regimen; Analysis of Lay Person Assessment Polarised Image; Test type: Superiority; p = 0.8887, ANOVA; ANOVA= average rate over all raters including effects of treatment and age stratum; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.12 to 0.14]
Statistical Analysis 3: Comparison: Test Product Regimen vs No Treatment Regimen; Analysis of Lay Person Assessment Non-Polarised Image; Test type: Superiority; p = 0.0224, ANOVA; ANOVA= average rate over all raters including effects of treatment and age stratum; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [0.02 to 0.28]
Statistical Analysis 4: Comparison: No Treatment Regimen vs Positive Control Regimen; Analysis of Lay Person Assessment Non-Polarised Image; Test type: Superiority; p = 0.8253, ANOVA; ANOVA= average rate over all raters including effects of treatment and age stratum; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.15 to 0.12]

5. Secondary Outcome: Change From Baseline in Evaluator's Assessment of Total Blemish Count at Week 1, 4, and 8
Description: A treatment blind, trained and qualified evaluator counted the total number of facial blemishes on the forehead, cheeks and chin of the participants.
Time Frame: At Baseline, Week 1, 4 and 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Total Blemish Count
Arm/Group | Test Product Regimen | No Treatment Regimen | Positive Control Regimen
Number analyzed (Participants) | 44 | 44 | 44
Total Blemish Count
  At Week 1: number analyzed (Participants) | 44 | 43 | 43
  At Week 1 | -0.70 (4.338) | -1.05 (3.331) | -0.93 (3.460)
  At Week 4: number analyzed (Participants) | 42 | 42 | 41
  At Week 4 | -3.86 (3.143) | -2.76 (4.154) | -4.00 (4.461)
  At Week 8: number analyzed (Participants) | 41 | 42 | 41
  At Week 8 | -5.68 (3.889) | -3.79 (3.626) | -5.12 (4.507)

6. Secondary Outcome: Change From Baseline in Sebumeter Values at Week 1, 4 and 8
Description: A treatment blinded, trained and qualified evaluator conducted instrumental measurements of skin sebum levels. Measurement of skin sebum levels was performed by with a Sebumeter SM 815. The measurement principle of the SM 815 is based on grease spot photometry. The translucent tape of the device is brought into contact with skin and becomes increasingly transparent in response to surface oil. The tape is inserted into the aperture of the device and its transparency measured by light transmission, with increased transmission signifying increased oiliness. The software outputs mass sebum levels as a function of area. Sebumeter measurements were taken in triplicate at the central forehead (above the eyebrows) with the participant lying horizontally, on their back.
Time Frame: At Baseline, Week 1, 4 and 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micrograms (μg)/square centimeter (cm^2)
Arm/Group | Test Product Regimen | No Treatment Regimen | Positive Control Regimen
Number analyzed (Participants) | 44 | 44 | 44
Micrograms (μg)/square centimeter (cm^2)
  At Week 1: number analyzed (Participants) | 44 | 43 | 43
  At Week 1 | -54.98 (133.157) | -70.50 (131.654) | -52.19 (116.797)
  At Week 4: number analyzed (Participants) | 42 | 42 | 41
  At Week 4 | -49.57 (128.821) | -67.52 (139.278) | -21.67 (114.170)
  At Week 8: number analyzed (Participants) | 41 | 42 | 41
  At Week 8 | -86.49 (118.708) | -87.04 (114.207) | -65.85 (111.936)

7. Secondary Outcome: Change From Baseline in Sebum Excretion Rate at Week 1, 4 and 8
Description: The forehead of each participant was thoroughly cleansed by the investigator or designee using cotton pads saturated with 70% Isopropyl Alcohol and, after 5 minutes, the central area of the forehead above the eyebrows was measured in triplicate with a Sebumeter. The same area was measured in triplicate 90 minutes after cleansing. The sebum excretion rate was calculated by the difference in 90th minutes and 5th minute Sebumeter values.
Time Frame: At Baseline, Week 1, 4 and 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μg/cm^2
Arm/Group | Test Product Regimen | No Treatment Regimen | Positive Control Regimen
Number analyzed (Participants) | 44 | 44 | 44
μg/cm^2
  At Week 1: number analyzed (Participants) | 44 | 43 | 43
  At Week 1 | 20.36 (135.959) | 38.72 (149.325) | 66.73 (161.570)
  At Week 4: number analyzed (Participants) | 42 | 42 | 41
  At Week 4 | 30.49 (153.074) | 44.97 (125.342) | 53.17 (137.181)
  At Week 8: number analyzed (Participants) | 41 | 42 | 41
  At Week 8 | 38.04 (162.934) | 32.91 (148.784) | 67.10 (112.039)

ADVERSE EVENTS:
Time Frame: Approximately 57 days
Description: 1 participant was misallocated to treatment (received "no treatment" instead of "positive control"). This means 45 participants were in safety population for "no treatment".However, per convention, ITT population is defined based on intended treatment allocation.While 1 subject incorrectly received "no treatment",they were initially allocated to "positive control". Therefore, this participant was included in ITT population for "positive control" but safety population for "no treatment".
Arm/Group | Test Product Regimen | No Treatment Regimen | Positive Control Regimen
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/45 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/45 | 0/43
Other Adverse Events (participants affected / at risk) | 1/44 | 2/45 | 5/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Product Regimen (N=44) | No Treatment Regimen (N=45) | Positive Control Regimen (N=43)
HEADACHE (Nervous system disorders) | 1 | 1 | 3
HYPERAESTHESIA (Nervous system disorders) | 0 | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 1
NASAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-05-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT03093181/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT03093181/SAP_001.pdf